CLINICAL TRIAL: NCT03452657
Title: Multicenter Clinical Study of Anti-VEGF Treatment on High Risk Diabetic Retinopathy (DR)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: RenJi Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Eye & ENT Hospital of Fudan University (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai 10th People's Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Xun Xu, Chief Physician, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLY201612
Record Dates: First submitted 2018-02-22; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Diabetic Retinopathy; Ranibizumab
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ranibizumab (Experimental): Participants received 0.5mg intravitreal ranibizumab injection
  Interventions: Drug: Ranibizumab
- Sham-injection (Sham Comparator): No drug involved in the sham procedure; patient's eye is anesthetized and a syringe without needle gently pressed on the conjunctival surface to simulate the force of an actual injection
  Interventions: Procedure: No drug

INTERVENTIONS:
Drug: Ranibizumab — Participants in arm Ranibizumab will receive ranibizumab injection every 4 weeks for the first 3 months, followed by re-injections every 3 months until 1year
  Other Names: Lucentis
  Arms: Ranibizumab
Procedure: No drug — Participants in arm Sham-injection will receive sham injection every 4 weeks for the first 3 months, followed by re-injections every 3 months until 1year.
  Arms: Sham-injection

SUMMARY:
The purpose of this study is to determine the efficacy and safety of intravitreous ranibizumab treatment versus sham injections for prevention of high-risk DR.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, multi-center, sham-controlled clinical trial. In this trial, 118 subjects will be enrolled. Subjects with signed informed consent are screened and assigned randomly (1:1) to one of the following parallel groups: Group A-Intravitreous 0.5 mg ranibizumab injections and Group B-sham injections. All participants have visits at 0 month, 1 month, and 2 months, followed by visits every 3 months thereafter through 1 year. The main efficacy and safety outcomes assessment will be finished at the end of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years;
2. Diagnosis of diabetes mellitus (type 1 or type 2);
3. The fundus color photography was graded by Reading Center as grade 47-53;
4. Patients have not received Pan Retinal Photocoagulation (PRP: laser spots on fundus outside hemal arch are less than 100);
5. HbA1C≤ 10%;
6. Media clarity and pupillary dilation sufficient to obtain adequate fundus examinations;
7. No central subfield macular edema.

Exclusion Criteria:

1. Ocular infection, including conjunctivitis, chalazion, or substantial blepharitis;
2. Proliferative diabetic retinopathy;
3. History of prior vitreous hemorrhage within 2 months;
4. An ocular condition is presented (other than DR), (e.g., retinal vein or artery occlusion, CNV, retinal detachment, macular hole, vitreomacular traction, etc.);
5. Evidence of iris neovascularization;
6. Evidence of uncontrolled glaucoma( Intraocular pressure >25 mmHg with glaucoma medication) or history of anti-glaucoma surgery;
7. Server cataract that influences judgment or needs cataract surgery in 6 months;
8. Aphakia;

   Received other ocular treatment:
9. History of intravitreal injection of corticosteroid within 3 months, or peribulbar injection of corticosteroid within 1 month;
10. History of vitreous surgery;
11. History of PRP ≥ 2 times or within 6 months in the study eye;
12. History of focal laser treatment within 3 months or laser treatment involving fovea ≥ 2 times in the past in the study eye;
13. History of anti-VEGF treatment within 6 months in the study eye or history of anti-VEGF treatment within 3 months in the non-study eye;
14. History of any intraocular surgery within 3 months;
15. History of macular surgery within 3 months;

    Have any following condition of systemic diseases:
16. Unsatisfactory blood glucose control within 3 months (defined as turn oral antidiabetic drugs into insulin therapy/insulin pump treatment or daily insulin injection times doubled);
17. Impaired renal function (Crea: 2 times higher than the upper limit of the normal laboratory center) or liver dysfunction (ALT, AST: 2 times higher than the upper limit of the normal laboratory center );
18. Poor blood pressure control (defined as systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 95 mmHg under antihypertensive therapy);
19. Any systemic infection that requires oral, intramuscular or intravenous administration ;
20. Stroke, transient ischemic attack, myocardial infarction or acute congestive heart failure occurred within 6 months before the screening;
21. Coagulation dysfunction (prothrombin time ≥ normal upper limit of 3 seconds, activated partial thromboplastin time ≥ normal upper limit of 10 seconds);
22. Drugs that are toxic to the lens, retina, or optic nerve are being used or may be required during the study (such as deferoxamine, chloroquine, hydroxychloroquine, tamoxifen, phenothiazine or ethambutol, etc.);
23. Have a diagnosis of systemic immune diseases (such as ankylosing spondylitis, systemic lupus erythematosus, etc.) or any uncontrollable clinical problems (such as AIDS, malignancy, active hepatitis, severe mental, neurological, cardiovascular, Respiratory and other diseases, etc.);
24. Known allergy to fluorescein dye, or protein products for treatment or diagnosis, or allergies to more than two drugs and / or nonpharmacological factors, or is suffering from allergic diseases;

    Other:
25. No use of effective contraception; Note: The following conditions are not excluded. I. Amenorrhea 12 months under natural circumstances, or natural amenorrhea for 6 months and serum follicle-stimulating hormone levels <40 mIU / ml; Ii. Bilateral ovariectomy with or without hysterectomy after 6 weeks; Iii. Use of one or more of the following acceptable contraceptive methods: sterilization (male with bilateral vasectomy, resection) , hormone contraceptive (implantable, patch-type, oral) , O IUD, or double barrier method; Iv. Reliable contraceptive measures used throughout the whole study period and adherence to the 30 days of discontinuation of the study drug (unacceptable contraceptive methods: regular abstinence - calendar, ovulation, body temperature, post-ovulation, Row fine);
26. Pregnant (pregnancy in this test is defined as urine pregnancy test positive) or lactating women;
27. Within 3 months (if the test drug has a long half-life and five half-life periods > 3 months, the time is 5 half-life periods) before screening, participated clinical trials of any drug (not including vitamins and minerals);
28. Those that researchers believe need to be excluded.

Exit Criteria:

During the clinical trial, patients may withdraw from the trial at any time for their own consideration or at the request of the investigator. For each subject who withdrawn from the trial, the investigator must detail the exit date, reasons, and other information in the case report form and original documents.

Subjects must withdraw from the study if:

1. Withdrawal of informed consent;
2. Participating in other clinical trials of new drugs during the trial;
3. Pregnancy during the trial;
4. Occurrence of ocular serious adverse events;
5. For safety, the researcher consider that the subject should withdraw from the trial.

Subjects may withdraw from the study early because of the following conditions:

1. Lost to follow-up;
2. Compliance issues;
3. Delay of injection more than 30 days for any reason;
4. Retinal laser photocoagulation is required during the trial;
5. Researchers consider that the treatments in this study (including remedial treatment) are no longer suitable for DME therapy in subjects;
6. Occurrence of adverse events or serious adverse events (subjects that need hospitalization or prolongation of hospital stay due to adverse events, without affecting the safety and efficacy evaluation, may not exit);
7. Use of prohibited drugs during the study;
8. Deviation from the research protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of eyes with a ≥ 2-step improvement in the ETDRS Diabetic Retinopathy Severity Scale (DRSS) score | 1 year
  Baseline ETDRS DRSS: None (level 10); Mild to moderate nonproliferative DR (levels 14, 15, 20, 35, and 43); Moderately severe/severe nonproliferative DR (levels 47 and 53); Mild/moderate/high-risk/advanced proliferative DR (levels 61, 65, 71,75, 81, and 85)

SECONDARY OUTCOMES:
Change from baseline in CRT (central retinal thickness) | 1 year
  Assessed on Optical Coherence Tomography (OCT)
Mean change from baseline in best-corrected visual acuity (BCVA) | 1 year
  Visual function of the study eye was assessed using the ETDRS protocol.
Proportion of eyes that meet the protocol-defined failure criteria | 1 year
  Failure criteria: Evidence of progression to PDR:
  1. Retinal neovascularization
  2. Iris neovascularization
  3. PDR related clinical manifestations: vitreous hemorrhage, tractive retinal detachment, etc..
  Patients who meet failure criteria will receive salvage therapy: PRP treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xun Xu, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (7):
- China (7):
  - Eye and ENT hospital of Fudan University, Shanghai
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai ninth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Sixth People's Hospital Affiliated to Shanghai Jiaotong University, Shanghai
  - Shanghai Tenth People's Hospital of Tongji University, Shanghai
  - Shanghai Tongji Hospital of Tongji University, Shanghai
  - Xinhua Hospital Afflilliated to Shanghai Jiaotong University School of Medicine, Shanghai